CLINICAL TRIAL: NCT02638441
Title: Psychological Profile of Women With Infertility in Egypt: A Comparative Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Bahaa El Din, lecturer, Ain Shams Maternity Hospital
Other Study IDs: ADin
Record Dates: First submitted 2015-12-15; First posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Infertility
Keywords: psychological health; women; anxiety; depression
MeSH Terms: conditions — Infertility; Psychological Well-Being; Anxiety Disorders; Depression | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: hospital anxiety and depression scale — Detection of infertility effect on emotional status
  Other Names: emotional distress of women with infertility

SUMMARY:
The aim of this study is to determine the prevalence of psychological affection in infertile egyptian women

DETAILED DESCRIPTION:
Comparative cross sectional study

ELIGIBILITY:
Inclusion Criteria:

Control group:

* Pregnant women.
* At least one live birth.
* Age group 20-40 years.

Clinical group:

* Infertile women either primary or secondary according to (WHO,2013).
* Age group 20-40ys.
* Different levels of education.
* Different methods of treatment of infertility (medical or IVF)
* Half of them from rural area the other half from urban area.

Exclusion Criteria:

* Male factor of infertility.
* The women with psychiatric disorders.
* The women with physical and medical disorders.
* The women whose current pregnancy has any problems (e.g. growth retardation, macrosomia, placenta previa, threatened abortion, or preterm labour).
* The women with history of intrauterine fetal death.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will be conducted at the department of Obstetrics and Gynecology of Ain shams university and Zagazig university and some private centres for the treatment of infertility. It will include 400 women, divided into two groups (control group and clinical group) starting from January 2016.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
determination of the prevalence of depression among infertile women | 6 months
  questionnaire will be used to collect qualititiative data from women

CONTACTS AND LOCATIONS:
Overall Officials: sherif a akl, Study Director — professor of obstetric and gynecology

IPD SHARING:
Plan to Share IPD: Yes